CLINICAL TRIAL: NCT01394913
Title: A Prospective, Double-blind, Randomized Study to Compare Efficacy of Two Etanercept Regimens (REUMATOCEPT® Versus ENBREL®) for Treatment of Rheumatoid Arthritis
Brief Title: Comparison of Two Etanercept Regimens (REUMATOCEPT® Versus ENBREL®) for Treatment of Rheumatoid Arthritis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ETAEMS0411
Record Dates: First submitted 2011-07-12; First posted 2011-07-15 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reumatocept 25mg (Experimental): 50mg each week for 30 weeks
  Interventions: Drug: Reumatocept (etanercept)
- Enbrel 25mg (Active Comparator): 50mg each week for 30 weeks
  Interventions: Drug: Enbrel (etanercept)

INTERVENTIONS:
Drug: Reumatocept (etanercept) — 50mg each week for 30 weeks
  Arms: Reumatocept 25mg
Drug: Enbrel (etanercept) — 50mg each week for 30 weeks
  Arms: Enbrel 25mg

SUMMARY:
This study is a comparison of safety and efficacy of two etanercept regimens (REUMATOCEPT® versus ENBREL®) for treatment of Rheumatoid Arthritis.

DETAILED DESCRIPTION:
Study design:

• Double blinded, non-inferiority, prospective parallel-group, intend to treat trial.

Study design:

* Experiment duration: 30 weeks
* 9 visits (days 0, 14, 42, 70, 98, 126, 154, 182, 210)
* Health Assessment Questionnaire (HAQ) evaluation
* Disease Activity Score (DAS28) evaluation
* Clinical Disease Activity Index (CDAI) evaluation
* American College of Rheumatology criteria (ACR) evaluation
* Visual Activity Schedule(VAS) evaluation
* Adverse events evaluation

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be able to understand the study procedures agree to participate and give written consent.
2. Patients with clinical diagnosis of moderate to severe rheumatoid arthritis according to American College of Rheumatology (ACR) criteria;
3. Patients with at least 6 swollen joints
4. Patients with partial response in treatment with methotrexate for 2 months

Exclusion Criteria:

1. Pregnancy and Lactation
2. Patients with uncontrolled hypertension
3. Patients with other rheumatic disease such as Sjogren syndrome, systemic lupus erythematosus or spondyloarthritis
4. Non-steroidal anti-inflammatory drug in the last 4 weeks
5. Any pathology or past medical condition that can interfere with this protocol
6. Patients with immunodeficiency and/or immunosuppressive disease;
7. Other conditions deemed reasonable by the medical investigator as to the disqualification of the individual from study participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2014-03 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy | day 1 to day 210
  1. Health Assessment Questionnaire (HAQ)
  2. Disease Activity Score (DAS28)
  3. Clinical Disease Activity Index (CDAI)
  4. American College of Rheumatology criteria (ACR)
  5. Visual Activity Schedule(VAS)

SECONDARY OUTCOMES:
Safety | day 1 to day 210
  Adverse events will be collected and followed in order to evaluate safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Pinho, MD, Study Director — EMS
Locations (1):
- Associação de Assitência à Criança Deficiente, São Paulo, Brazil